CLINICAL TRIAL: NCT05490953
Title: Enhancing Effect on Tumour Apoptosis With the Combined Use of Pentoxifylline Plus Chemotherapeutical Agents in Pediatrics and AYA Patients With Hodgkin´s Lymphoma
Brief Title: Enhancing Effect on Tumour Apoptosis With the Use of Pentoxifylline in Patients With Hodgkin Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Ramón Óscar González-Ramella, Ph.D, Titular Research Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI-03122
Record Dates: First submitted 2022-06-29; First posted 2022-08-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; Pentoxifylline; Apoptosis; Pediatric and adolescent and young adult patients
MeSH Terms: conditions — Hodgkin Disease | interventions — Pentoxifylline

STUDY DESIGN:
Intervention Model Description: Patients who agree to participate in this study, by signing the consent and/or informed assent, will be randomly assigned to each of the two study groups: Group A: Patients with conventional treatment based on the OEPA/COPDAC, ABVD or BEACOPP scheme plus placebo, during the first two cycles of chemotherapy. Group B: patients with conventional treatment based on the OEPA/COPDAC, ABVD or BEACOPP scheme plus pentoxifylline, during the first two cycles of chemotherapy.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be stratified at randomization based on their clinical stage at diagnosis, according to the Cotswold classification system, into limited-stage (stage I or II disease without B symptoms and absence of bulky or stage IB disease without bulky disease) and advanced stage (patients with stage II disease with B symptoms or bulky disease, or stage III or IV disease). In addition, a random permutation method with blocks of size 6 will be used, thus creating 5 blocks of size 6 patients each. Each patient will be classified into a specific study group (Group A: conventional treatment plus placebo; group B: conventional treatment plus pentoxifylline).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A with placebo (Placebo Comparator): Patients with conventional treatment based on the OEPA/COPDAC, ABVD or BEACOPP scheme plus placebo, during the first two cycles of chemotherapy.
  Interventions: Drug: Placebo
- Group B with pentoxifylline (Experimental): Patients with conventional treatment based on the OEPA/COPDAC, ABVD or BEACOPP scheme plus pentoxifylline, during the first two cycles of chemotherapy.
  Pentoxifylline dose of 20 mg/kg/day, maximum dose 1200 mg/day
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Patients will be treated pentoxifylline during the first two chemotherapy cycles of their respective treatment.
  Other Names: Experimental Group
  Arms: Group B with pentoxifylline
Drug: Placebo — Patients will be treated with placebo during the first two chemotherapy cycles of their respective treatment.
  Other Names: Placebo Group
  Arms: Group A with placebo

SUMMARY:
Hodgkin's Lymphoma (HL) is a neoplasm that affects the lymph nodes and the lymphatic system. In Mexico, HL is the seventh most incident cancer and the ninth with the highest mortality. It is characterized by the presence of Reed-Sternberg (HRS) cells derived from B cells of the germinal center. They harbor mutations that activate the NF-κB pathway, favoring cell survival and their reprogramming. Currently, the available therapeutic options are chemotherapy and radiotherapy, achieving cure rates of 75% in patients in advanced stages, in which 70% of these are found at the time of diagnosis. The investigators proposed the use of pentoxifylline (PTX) as a therapeutic option to enhance the antitumor effect generated by the treatment since it can increase the efficacy of apoptosis, in vitro and in vivo, induced by doxorubicin, cisplatin, and adriamycin in human leukemic and cervical cancer cells, through inhibition of NF-κB by preventing phosphorylation of serine 32 of the inhibitor κB; it also decreases the expression of Bcl-2 and Bcl-XL, induces the releasement of cytochrome c and caspases 3, 9, and cleavage of caspase 8. The investigators evaluated the effects of PTX during the steroid window phase at induction to remission in pediatric patients with LLA of a recent diagnosis, where it was shown that the combined treatment of prednisone (PRD) with PTX achieves greater percentages of apoptosis compared to individual treatment. In addition, the effect of PTX on the expression of genes associated with apoptosis was evaluated; where it was shown that it activates the intrinsic and extrinsic pathways of apoptosis. Fortilin is a protein whose serum levels increase 2.4 times more after treatment with chemotherapy or radiotherapy in patients with malignancies, so it is considered a specific and sensitive biomarker of early apoptosis in vivo. The present protocol will evaluate the enhancing effect of PTX on tumor apoptosis in combination with chemotherapeutical agents in pediatric and AYA patients with HL. Apoptosis will be measured in vivo by quantifying serum levels of fortilin and cytochrome c in participants before and after treatment by ELISA; as well as an evaluation of the clinical response based on the results of the PET-Scan, overall and event-free survival according to the Kaplan-Meier curves, and the adverse effects associated with the use of PTX according to the common terminology criteria for adverse events and causality algorithms.

DETAILED DESCRIPTION:
Hodgkin Lymphoma (HL) is a B-cell-derived neoplasm that involves the lymph nodes and lymphatic system. In Mexico, HL is seventh cancer with the highest incident rates and the ninth with the highest mortality.

The incidence of this pathology has a bimodal distribution, with the first peak of appearance among adolescents and young adults within an age range that goes from 15 to 35 years, followed by a second peak in adults 55 years of age and older.

This neoplasm is characterized by the presence of Reed-Sternberg cells (HRS), which are distinguished by being large with multinucleate or bilobed nuclei and being derived from B lymphocytes of the germinal center. They have a partial loss of the B phenotype and classical lineage markers. They harbor mutations that activate the NF-κB pathway, which regulates antiapoptotic factors, the expression of proinflammatory cytokines, and the reprogramming of B cells.

Patients with HL frequently present asymptomatic, painless, and slowly progressive lymphadenopathy. There may also be systemic symptoms such as B symptoms which are defined by the presence of deep night sweats, unexplained weight loss of >10% of total body weight within the previous 6 months at diagnosis, and persistent or recurrent fever ≥38˚C.

Excisional biopsy of potentially involved lymph nodes is the gold standard for establishing the diagnosis of HL. A histopathological study is performed, in which the presence of diagnostic HRS cells must be found in an adequate microenvironment and the expression of CD30 and CD15.

Treatment is implemented based on the stage of the disease, with limited stages being an initial phase with chemotherapy followed by a consolidation phase with or without targeted radiotherapy. In limited favorable stages, it is recommended to apply 2 to 3 cycles of chemotherapy or 4 cycles for those with limited unfavorable stages. The scheme with the best cure rates is ABVD (adriamycin or doxorubicin, bleomycin, vinblastine, and dacarbazine). For advanced disease, the application of 6 cycles of combined chemotherapy using the BEACOPP scheme (bleomycin, etoposide, doxorubicin or adriamycin, cyclophosphamide, vincristine, procarbazine, and prednisone).

Pentoxifylline (PTX) is a non-specific phosphodiesterase inhibitor belonging to the methylxanthine family. It has been reported that PTX can increase the efficacy of certain antitumor drugs through the inhibition of NF-κB. This can prevent the phosphorylation of serine 32 of the inhibitor of NF-κB (I-κB), thus preventing the activity of NF-κB and being able to activate certain proapoptotic genes. In addition, PTX is capable of sensitizing multidrug-resistant cells by down-regulating P-glycoprotein.

The efficacy of PTX has been reported, both in vitro and in vivo, in increasing apoptosis induced by some chemotherapeutic drugs such as doxorubicin, cisplatin, and adriamycin, both in humans leukemia cells and in cervical cancer cells and an increase in survival in murine models of lymphoma. It has also been shown that PTX decreases the expression of Bcl-2 and Bcl-XL. They also induce the release of cytochrome C and caspases 3, 9 and cleavage of caspase 8, resulting in increased apoptosis in the human leukemia cell line U937.

PTX also manages to significantly inhibit cellular senescence, a state that is induced by chemotherapy, which, although characterized by the non-replication of cells, continues to be alive, facilitating tumor growth.

Fortilin is a 172-amino acid protein that can be found in the cytosol, nucleus, extracellular space, mitochondria, and peripheral blood. In 2010, I. Sirois et al. identified the presence of fortilin as the most abundant protein in nanovesicles secreted by apoptotic cells. In addition, it was possible to demonstrate one of the extracellular functions of fortilin in the context of apoptosis, since these nanovesicles secreted by apoptotic cells were able to induce an antiapoptotic phenotype regardless of the cell type in question.

In a study conducted by Sinthujaroen et al., the potential use of serum fortilin as a peripheral biomarker associated with apoptosis was evaluated. Fortilin was shown to be present in the peripheral blood of healthy participants and patients with solid malignant tumors. In those patients without malignancies, the mean values were 75.57 ± 45.79 ng/mL with no significant difference between sex or age. Likewise, serum levels of this were measured in cancer patients before and after the administration of chemotherapy drugs or radiotherapy, and a 2.4-fold increase in their serum levels was observed after treatment.

Serum fortilin was considered a unique biomarker of apoptosis in vivo, thus, it is correlated that high serum levels are associated with greater tumour apoptosis.

Within the background that gave rise to this study, a pilot study was carried out where the effects of the use of PTX during the steroid window on the induction of remission in pediatric patients with a recent diagnosis of acute lymphocytic leukemia (ALL) were evaluated. For this study, patients were classified into 3 groups: Group 1 treated with prednisone (PRD) alone, Group 2 treated with a combination of PRD/PTX, and Group 3 with healthy control.

Significant differences were observed in the rate of apoptosis after treatment between the groups treated only with PRD and those treated together with PTX, with a higher percentage observed in group 2 treated with PTX (PTX 16.5±6.04% vs. PRD 9.2± 3.1; p=<0.001). In addition, it was shown that the combined treatment of PRD with PTX gives higher percentages of apoptosis in leukemic cells compared to individual treatment with PRD, showing that PTX can increase glucocorticoid-induced cell death in pediatric patients with ALL.

In this same group of patients, the effect of PTX on the expression of genes associated with apoptosis was evaluated. A significant difference between the number of genes that are regulated, both up and down, when PTX is added compared to treatment with PRD alone was evidenced.

Among the genes that were modified in their expression by the PTX/PRD treatment, were those associated with FOXO3A, TNF receptors, DISC-associated genes such as FADD, and caspase-8 and -10 genes. The genes found to be downregulated were associated with BCL-2, the NF-κB pathway, and CDKN2A. However, there was also downregulation of proapoptotic genes (JUN, LTA, AKT, TRAF3, and PMAIP1) and upregulation of some antiapoptotic (BRIC3 and CFLAR).

Cancer is one of the leading causes of morbidity and mortality in children and adolescents around the world. In Mexico, is considered one of the biggest public health problems in pediatric patients since it represents the first cause of death in this age group.

HL comprises 6% of all childhood cancers. Although cure rates of up to 90-95% are currently reported in early stages, only 30% of patients are found in these stages at the time of diagnosis, leaving a large percentage of patients in advanced stages at diagnosis. For this latter group, currently available treatments have only achieved cure rates of approximately 75% of cases.

In addition, the therapeutic options are based on chemotherapeutic drugs and radiotherapy, which have repercussions on patients both in short and long term. Among the main associated adverse effects are cardiomyopathies, coronary heart disease, pulmonary toxicity, and the development of secondary neoplasms, both hematological and solid tumors; these constitute one of the main causes of mortality in long-term survivors.

Based on the antitumor effects of PTX and part of the pathophysiology of HL, the administration of PTX in combination with the drugs used in the standard chemotherapy scheme for the treatment of HL is proposed as a pharmacological strategy to increase the rate of apoptosis in lymphoma cells during the treatment of pediatric and adolescent/young adult patients with newly diagnosed HL.

This way, it is expected that the increase in cell death will have a positive impact on the clinical response and both global and event-free survival of patients, in addition, to giving rise to future research where this drug is used in conjunction with current treatments for different hematological neoplasms such as non-Hodgkin lymphoma.

The investigators hypothesize that pentoxifylline, when used in conjunction with chemotherapeutic agents, manages to enhance the effect that the latter has in inducing tumor cell apoptosis in vitro and in patients with Hodgkin lymphoma, which leads to an improvement in survival, and their clinical response.

The aim of the study is to evaluate the potentiating effect on cell apoptosis generated by the combined use of pentoxifylline with chemotherapeutic agents in patients with Hodgkin lymphoma during pharmacological treatment.

The universe of study will be pediatric, adolescent, and young adults patients with a recent diagnosis of Hodgkin lymphoma without prior treatment, from Pediatric Oncology and Hematology Service of the Hospital Civil de Guadalajara Dr. Juan I. Menchaca, and the Hospital Civil de Guadalajara Fray Antonio Alcalde in the Adult Hematology Service.

The sample size was evaluated based on the sample size formula for a given proportion, considering the proportion obtained in the protocol "Very early remission and increased apoptosis with the use of pentoxifylline in children with lymphoblastic leukemia acute" (Salceda Rivera et al., 2020).

To achieve statistically significant results a sample size of 30 patients was obtained, considering a proportion of 99%. Patients will be classified into two study groups: Group A: Patients with conventional treatment based on the OEPA/COPDAC, ABVD, or BEACOPP chemotherapy scheme plus placebo, during the first two cycles of chemotherapy. Group B: patients with conventional treatment based on the OEPA/COPDAC, ABVD, or BEACOPP chemotherapy scheme plus pentoxifylline, during the first two cycles of chemotherapy.

The dose of pentoxifylline is 20 mg/kg/day (maximum dose of 1200 mg), which will be indicated orally, without chewing or crushing, preferably accompanied by food. It will be administered one hour before the rest of the drugs that are part of the respective chemotherapy regimen.

Three peripheral venous blood samples will be obtained from the patients before the start of treatment (day 0), at the end of the first cycle of chemotherapy (day 30), and at the end of the second cycle (day 60). Plasma levels of indirect biomarkers of apoptosis (fortilin and cytochrome c) will be determined by ELISA; the results will be represented as the mean ± standard deviation in pg/mL.

The clinical response will be evaluated comparatively based on the physical examination and the data provided by the clinical file. Likewise, a positron emission tomography (PET) or Computed Axial Tomography will be performed at the time of diagnosis (day 0) and the end of the second cycle of chemotherapy (day 60). Event-free survival will be assessed using the Kaplan-Meier log-rank test.

Finally, the adverse effects will be determined according to the Common Terminology Criteria for Adverse Events. In addition, it will be determined if the presence of an adverse effect is correlated to the use of pentoxifylline using Karch & Lasagna, Naranjo, and FDA causality algorithms for adverse drug reactions.

The data will be represented as the mean ± the standard deviation of the values obtained. The data obtained will be analyzed by inferential statistics using the Mann-Whitney U test for parametric data. For qualitative variables, contingency tables will be used, to use squared Xi, in addition to multiple linear regression since multi variables will be used. The kappa (k) statistical test will be used to measure the strength of agreement between the causality algorithms. A statistically significant difference between the data will be considered when the p-value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and AYA (adolescents and young adults) patients (age up to 35 years of either sex) newly diagnosed with Hodgkin lymphoma regardless of clinical stage.
* Patients with the ability to swallow tablets.
* Patients who agree to enter the protocol by signing the informed consent personally or by the parent/guardian

Exclusion Criteria:

* Patients previously treated with chemotherapy, corticoids, and/or radiotherapy
* History of active acid peptic disease or gastrointestinal bleeding Intolerance to pentoxifylline and in general to xanthines
* Patients under treatment with anticoagulants, cimetidine, ciprofloxacin or theophylline
* Patients with severe bleeding, retinal hemorrhage or bleeding diathesis
* Serious cardiac arrhythmias (E.g. paroxysmal supraventricular tachycardia, congenital AV block, arrhythmias associated with congenital heart disease, digitalis poisoning, postoperative cardiac surgery, hypoxia, hypercapnia, electrolyte disturbances)
* Patients with hypotension
* Severe liver failure
* Moderate to severe renal insufficiency (with a glomerular filtration rate ≤ 30 mL/min)
* Patients admitted to the Intensive Care Unit at diagnosis
* Patients with treatment adherence of less than 80%
* Patients who wish to withdraw from the study or withdraw informed consent
* Patients who present grade III adverse events related to the drug under study
* Patients who become pregnant during the study

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral apoptosis (Fortilin) | At the end of the second cycle of chemotherapy (day 60 after starting chemotherapy, since each cycle of treatment is 30 days)
  3 samples of peripheral venous blood will be obtained from the patients from both study groups before the beginning of treatment (day 0), at the end of the first cycle of chemotherapy (day 30), and the end of the second cycle (day 60). Fortilin plasma levels will be determined using the translationally controlled human tumor protein ELISA kit (TPT1), according to the manufacturer's specifications. The optical density will be determined using a Biotek Synergy™ HT plate reader at a wavelength of 450nm. The results will be presented as the mean ± standard deviation in pg/mL.
  In the 3 blood samples that will be taken from the participants, the same marker will be evaluated. As it is the same variable, it will be measured with the same unit of measure (pg/mL) for the 3 blood samples.
  At the end of the study, it will be evaluated if there was any change in the plasma levels of fortilin (in pg/mL), either an increase or a decrease.
Peripheral apoptosis (Cytochrome c) | At the end of the second cycle of chemotherapy (day 60 after starting chemotherapy, since each cycle of treatment is 30 days)
  3 samples of peripheral venous blood will be obtained from the patients from both study groups before the beginning of treatment (day 0), at the end of the first cycle of chemotherapy (day 30), and the end of the second cycle (day 60). Cytochrome c plasma levels will be determined using the human cytochrome c ELISA kit, according to the manufacturer's specifications. The optical density will be determined using a Biotek Synergy™ HT plate reader at a wavelength of 450nm. The results will be presented as the mean ± standard deviation in pg/mL.
  In the 3 blood samples that will be taken from the participants, the same marker will be evaluated. As it is the same variable, it will be measured with the same unit of measure (pg/mL) for the 3 blood samples.
  At the end of the study, it will be evaluated if there was any change in the plasma levels of fortilin (in pg/mL), either an increase or a decrease.

SECONDARY OUTCOMES:
Assessment of the clinical response by positron emission tomography (PET) | At the end of the second cycle of chemotherapy (day 60 after starting chemotherapy, since each cycle of treatment is 30 days)
  The clinical response will be comparatively evaluated by PET at the time of diagnosis and at the end of the treatment scheme (day 60 after starting chemotherapy, since each treatment cycle is 30 days). The change in tumor masses will be objectively compared by evaluating the PETs with the Deauville criteria, a 5-point scale:
  * 1 to 3 points: Negative, achieving a positive clinical response.
  * 4 to 5 points: Positive, with a negative clinical response.
Assessment of the clinical response by Computerized Axial Tomography | At the end of the second cycle of chemotherapy (day 60 after starting chemotherapy, since each cycle of treatment is 30 days)
  In case it is not possible to have access to perform PET to the participants, the clinical response will be evaluated comparatively using Computerized Axial Tomography at the time of diagnosis, and at the end of the treatment scheme (day 60 after starting chemotherapy, since each cycle of treatment is 30 days). The change in tumor masses will be subjectively compared to determine if there was a clinical response:
  * Presence of clinical response: Absence of previously identified tumor masses or a decrease in their size.
  * No presence of clinical response: Persistence of previously identified tumor masses or increase in their size, as well as the presence of new tumor masses.
Assessment of the clinical response | At the end of the second cycle of chemotherapy (day 60 after starting chemotherapy, since each cycle of treatment is 30 days)
  The clinical response will be evaluated comparatively based on the physical examination and the data provided by the medical file. Likewise, a positron emission tomography (PET) or Computerized Axial Tomography will be performed at the time of diagnosis, after the second cycle of chemotherapy, and at the end of the treatment scheme. The change of the tumour masses will be objectively compared or the results will be interpreted based on the Deauville criteria.
Determination of event-free survival | A 24-month follow-up will be given after completion of the corresponding treatment, at the time, survival will be evaluated.
  The event-free survival will be assessed using the Kaplan-Meier log-rank test, considering a statistically significant difference when a p-value less than 0.05 is obtained
Assessment of the severity of adverse effects | A 24-month follow-up will be given after finishing the corresponding treatment, at that time, the adverse effects will be studied.
  The severity of the adverse effects that patients may experience associated with the use of pentoxifylline will be determined according to the Common Terminology Criteria for Adverse Events (CTCAE), classifying them in grades from 1 to 5:
  * Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL: preparing meals, shopping for groceries or clothes, using the telephone, etc.)
  * Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL (bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden)
  * Grade 4: Life-threatening consequences; urgent intervention indicated.
  * Grade 5: Death related to adverse effects.
Correlation of adverse effects with pentoxifylline | A 24-month follow-up will be given after finishing the corresponding treatment, at that time, the adverse effects will be studied.
  To determine if the presence of an adverse effect is correlated to the use of pentoxifylline and not to the effects related to the rest of the chemotherapeutic drugs or due to symptoms associated with the pathology, the causality algorithms of Karch & Lasagna, Naranjo, and the FDA for adverse drug reactions will be used. The correlation is classified as:
  * Definitive
  * Likely
  * Possible
  * Unlikely

CONTACTS AND LOCATIONS:
Overall Officials: Ramón O. González Ramella, PhD, Study Director — University of Guadalajara
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
It's not contemplated to share the data of the participants since it is personal information. During the development of the study, the anonymity of the participants will be maintained at all times, protecting their security and identity.

REFERENCES:
- [Background] Wang HW, Balakrishna JP, Pittaluga S, Jaffe ES. Diagnosis of Hodgkin lymphoma in the modern era. Br J Haematol. 2019 Jan;184(1):45-59. doi: 10.1111/bjh.15614. Epub 2018 Nov 8. PMID 30407610
- [Background] Connors JM, Cozen W, Steidl C, Carbone A, Hoppe RT, Flechtner HH, Bartlett NL. Hodgkin lymphoma. Nat Rev Dis Primers. 2020 Jul 23;6(1):61. doi: 10.1038/s41572-020-0189-6. PMID 32703953
- [Background] Weniger MA, Kuppers R. Molecular biology of Hodgkin lymphoma. Leukemia. 2021 Apr;35(4):968-981. doi: 10.1038/s41375-021-01204-6. Epub 2021 Mar 8. PMID 33686198
- [Background] Mathas S, Hartmann S, Kuppers R. Hodgkin lymphoma: Pathology and biology. Semin Hematol. 2016 Jul;53(3):139-47. doi: 10.1053/j.seminhematol.2016.05.007. Epub 2016 May 13. PMID 27496304
- [Background] Hernandez-Flores G, Ortiz-Lazareno PC, Lerma-Diaz JM, Dominguez-Rodriguez JR, Jave-Suarez LF, Aguilar-Lemarroy Adel C, de Celis-Carrillo R, del Toro-Arreola S, Castellanos-Esparza YC, Bravo-Cuellar A. Pentoxifylline sensitizes human cervical tumor cells to cisplatin-induced apoptosis by suppressing NF-kappa B and decreased cell senescence. BMC Cancer. 2011 Nov 10;11:483. doi: 10.1186/1471-2407-11-483. PMID 22074157
- [Background] Bravo-Cuellar A, Ortiz-Lazareno PC, Lerma-Diaz JM, Dominguez-Rodriguez JR, Jave-Suarez LF, Aguilar-Lemarroy A, del Toro-Arreola S, de Celis-Carrillo R, Sahagun-Flores JE, de Alba-Garcia JE, Hernandez-Flores G. Sensitization of cervix cancer cells to Adriamycin by Pentoxifylline induces an increase in apoptosis and decrease senescence. Mol Cancer. 2010 May 19;9:114. doi: 10.1186/1476-4598-9-114. PMID 20482878
- [Background] Lerma-Diaz JM, Hernandez-Flores G, Dominguez-Rodriguez JR, Ortiz-Lazareno PC, Gomez-Contreras P, Cervantes-Munguia R, Scott-Algara D, Aguilar-Lemarroy A, Jave-Suarez LF, Bravo-Cuellar A. In vivo and in vitro sensitization of leukemic cells to adriamycin-induced apoptosis by pentoxifylline. Involvement of caspase cascades and IkappaBalpha phosphorylation. Immunol Lett. 2006 Mar 15;103(2):149-58. doi: 10.1016/j.imlet.2005.10.019. Epub 2005 Nov 18. PMID 16388856
- [Background] Bravo-Cuellar A, Hernandez-Flores G, Lerma-Diaz JM, Dominguez-Rodriguez JR, Jave-Suarez LF, De Celis-Carrillo R, Aguilar-Lemarroy A, Gomez-Lomeli P, Ortiz-Lazareno PC. Pentoxifylline and the proteasome inhibitor MG132 induce apoptosis in human leukemia U937 cells through a decrease in the expression of Bcl-2 and Bcl-XL and phosphorylation of p65. J Biomed Sci. 2013 Feb 28;20(1):13. doi: 10.1186/1423-0127-20-13. PMID 23445492
- [Background] Gonzalez-Ramella O, Ortiz-Lazareno PC, Jimenez-Lopez X, Gallegos-Castorena S, Hernandez-Flores G, Medina-Barajas F, Meza-Arroyo J, Jave-Suarez LF, Lerma-Diaz JM, Sanchez-Zubieta F, Bravo-Cuellar A. Pentoxifylline during steroid window phase at induction to remission increases apoptosis in childhood with acute lymphoblastic leukemia. Clin Transl Oncol. 2016 Apr;18(4):369-74. doi: 10.1007/s12094-015-1376-x. Epub 2015 Sep 2. PMID 26329293
- [Background] Meza-Arroyo J, Bravo-Cuellar A, Jave-Suarez LF, Hernandez-Flores G, Ortiz-Lazareno P, Aguilar-Lemarroy A, Padilla-Corona M, Sanchez-Zubieta F, Gonzalez-Ramella O. Pentoxifylline Added to Steroid Window Treatment Phase Modified Apoptotic Gene Expression in Pediatric Patients With Acute Lymphoblastic Leukemia. J Pediatr Hematol Oncol. 2018 Jul;40(5):360-367. doi: 10.1097/MPH.0000000000001152. PMID 29683943
- [Background] Sinthujaroen P, Wanachottrakul N, Pinkaew D, Petersen JR, Phongdara A, Sheffield-Moore M, Fujise K. Elevation of serum fortilin levels is specific for apoptosis and signifies cell death in vivo. BBA Clin. 2014 Dec 1;2:103-111. doi: 10.1016/j.bbacli.2014.10.002. PMID 25558447
- [Background] Kuppers R. The biology of Hodgkin's lymphoma. Nat Rev Cancer. 2009 Jan;9(1):15-27. doi: 10.1038/nrc2542. Epub 2008 Dec 11. PMID 19078975
- [Background] Weniger MA, Kuppers R. NF-kappaB deregulation in Hodgkin lymphoma. Semin Cancer Biol. 2016 Aug;39:32-9. doi: 10.1016/j.semcancer.2016.05.001. Epub 2016 May 21. PMID 27221964
- [Background] Schwarzer R, Jundt F. Notch and NF-kappaB signaling pathways in the biology of classical Hodgkin lymphoma. Curr Mol Med. 2011 Apr;11(3):236-45. doi: 10.2174/156652411795243423. PMID 21375490
- [Background] de Oliveira KA, Kaergel E, Heinig M, Fontaine JF, Patone G, Muro EM, Mathas S, Hummel M, Andrade-Navarro MA, Hubner N, Scheidereit C. A roadmap of constitutive NF-kappaB activity in Hodgkin lymphoma: Dominant roles of p50 and p52 revealed by genome-wide analyses. Genome Med. 2016 Mar 17;8(1):28. doi: 10.1186/s13073-016-0280-5. PMID 26988706
- [Background] Hinz M, Lemke P, Anagnostopoulos I, Hacker C, Krappmann D, Mathas S, Dorken B, Zenke M, Stein H, Scheidereit C. Nuclear factor kappaB-dependent gene expression profiling of Hodgkin's disease tumor cells, pathogenetic significance, and link to constitutive signal transducer and activator of transcription 5a activity. J Exp Med. 2002 Sep 2;196(5):605-17. doi: 10.1084/jem.20020062. PMID 12208876
- [Background] Hernandez-Flores G, Bravo-Cuellar A, Aguilar-Luna JC, Lerma-Diaz JM, Barba-Barajas M, Orbach-Arbouys S. [In vitro induction of apoptosis in acute myelogenous and lymphoblastic leukemia cells by adriamycine is increased by pentoxifylline]. Presse Med. 2010 Dec;39(12):1330-1. doi: 10.1016/j.lpm.2010.07.013. No abstract available. French. PMID 20888731
- [Background] Sirois I, Raymond MA, Brassard N, Cailhier JF, Fedjaev M, Hamelin K, Londono I, Bendayan M, Pshezhetsky AV, Hebert MJ. Caspase-3-dependent export of TCTP: a novel pathway for antiapoptotic intercellular communication. Cell Death Differ. 2011 Mar;18(3):549-62. doi: 10.1038/cdd.2010.126. Epub 2010 Oct 22. PMID 20966960